CLINICAL TRIAL: NCT01615900
Title: Randomized Open Label Study Evaluating the Coverage by Teleconsultation Versus Standard Follow-up of Renal Transplant Patients According to a Risk Score of Early Graft Failure (KTFS)
Acronym: TELEGRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRD/11/06-O
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Renal Transplant Patient
Keywords: Renal graft; Teleconsultation; Kidney transplant failure score
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teleconsultation (Other)
  Interventions: Other: Teleconsultation / Standard consultation
- Standard consultation (Other)
  Interventions: Other: Teleconsultation / Standard consultation

INTERVENTIONS:
Other: Teleconsultation / Standard consultation — Stage 1: randomization. Two arms: teleconsultation and standard consultation
  Stage 2: calculation of Kidney Transplant Failure Score which will determine 4 sub-groups: teleconsultation high risk, teleconsultation low risk, standard consultation high risk and standard consultation low risk.
  Stage 3: follow-up (2 years) according to the group:
  * Standard consultation low risk: consultation every 2 months during one year and then every 3 months during one year
  * Standard consultation high risk: consultation every 6 weeks during one year and then every 2 months during one year
  * Teleconsultation low risk: same follow-up as "standard consultation low risk" group but all the consultations are teleconsultations
  * Teleconsultation high risk: same follow-up as "standard consultation high risk" group but the follow-up will be intensified by the addition of an intermediate teleconsultation (between 2 consultations)

SUMMARY:
The main objective of this study is to optimize the coverage of renal transplant patients thanks to a personalized follow-up based on a risk score of early graft failure (KTFS, Kidney Transplant Failure Score), associated with teleconsultations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Having received a deceased donor renal transplant one year ago
* Having an access internet high-speed
* Having a compatible computer and supporting the videoconference
* Calculable KTFS (Kidney Transplant Failure Score)
* Patient having participated in a therapeutic educational program
* Patient has given informed consent
* Patient insured

Exclusion Criteria:

* Patient under age 18
* Patient having received a multi-organ transplant (heart kidney / liver kidney / kidney pancreas / lung kidney / heart lung kidney)
* Patient non-compliant
* BK virus nephropathy or BK positive viremia
* CMV positive viremia
* Identified and treated psychiatric disorders
* Participation in another clinical study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events | 2 years
  The main objective of this study is to optimize the coverage of renal transplant patients thanks to a personalized follow-up based on a risk score of early graft failure (KTFS, Kidney Transplant Failure Score), associated with teleconsultations.

SECONDARY OUTCOMES:
Cost-effectiveness of the personalized follow-up | 2 years
Quality of life linked to the health of transplant patients | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France